CLINICAL TRIAL: NCT07336329
Title: Effectiveness of Periodic Use of Continuous Glucose Monitoring After Three Months of Continuous Use in Patients With Non-Insulin-Treated Type 2 Diabetes Patients: A Multicenter, Randomized, Parallel-Group, Open-Label, Non-Inferiority, Investigator-Initiated Trial
Brief Title: Continuous Glucose Monitoring in Non-Insulin Treated Type 2 Diabetes: Continuous vs. Periodic Use
Acronym: PERIODIC-CGM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Sun Joon, Moon, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBSMC 2025-07-031
Record Dates: First submitted 2026-01-10; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a non-inferiority trial comparing periodic versus continuous use of CGM
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Periodic CGM Use (Experimental): All participants first wear FreeStyle Libre 2 CGM continuously for 12 weeks to establish baseline glucose patterns. Only those with at least 50% sensor active time proceed to randomization. After randomization, participants in this arm wear CGM intermittently for 2 weeks at weeks 2, 6, and 10 (±3 days each). Each sensor is worn for 14 days then removed. During non-wearing periods, no CGM is used. Participants receive education on diet adjustment based on postprandial glucose from CGM. Existing diabetes medications are maintained without changes throughout the study.
  Interventions: Device: FreeStyle Libre 2 Continuous Glucose Monitoring
- Continuous CGM Use (Active Comparator): All participants first wear FreeStyle Libre 2 CGM continuously for 12 weeks to establish baseline glucose patterns. Only those with at least 50% sensor active time proceed to randomization. After randomization, participants in this arm continue to wear CGM continuously for 12 weeks with sensor replacement every 14 days (total 6 replacements). Participants receive education on diet adjustment based on postprandial glucose from CGM. Existing diabetes medications are maintained without changes throughout the study.
  Interventions: Device: FreeStyle Libre 2 Continuous Glucose Monitoring

INTERVENTIONS:
Device: FreeStyle Libre 2 Continuous Glucose Monitoring — FreeStyle Libre 2 continuous glucose monitoring system consisting of a sensor worn on the upper arm that measures interstitial glucose levels continuously for up to 14 days. Data is transmitted to a smartphone app (FreeStyle LibreLink). The sensor is a Class 3 medical device approved by MFDS (Korea). Participants receive education on adjusting diet based on postprandial glucose patterns observed through CGM. Existing diabetes medications (oral agents and/or GLP-1 agonists) are maintained without changes throughout the intervention period.

SUMMARY:
The goal of this clinical trial is to test whether wearing a continuous glucose monitor (CGM) part-time works as well as wearing it full-time in adults with type 2 diabetes who do not use insulin. The main questions it aims to answer are:

* Does wearing CGM part-time (2 weeks per month) control blood sugar as well as wearing it continuously?
* How do the two wearing patterns compare for blood sugar levels throughout the day, weight, blood pressure, and patient satisfaction?

Researchers will compare part-time CGM use to continuous CGM use to see if part-time use is just as effective for blood sugar control.

All participants will:

* Wear a CGM device continuously for 3 months to learn how their blood sugar responds to different foods and activities
* Then be randomly assigned to wear CGM either part-time (2 weeks each month) or continuously for another 3 months
* Replace the CGM sensor on their arm every 2 weeks
* Use a smartphone app to track their blood sugar readings
* Visit the clinic 3 times for blood tests and check-ups
* Receive education on adjusting diet based on their CGM readings
* Keep their current diabetes medications unchanged during the study

The study will last about 6 months total. Participants will use the FreeStyle Libre 2 CGM device, which is already approved for use in people with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 80 years at the time of informed consent
* Adults with type 2 diabetes not using insulin
* Patients treated with GLP-1 agonist, oral hypoglycemic agents, and/or lifestyle modifications
* Patients who have maintained stable diabetes treatment for at least 3 months without changes
* HbA1c between 7.5% and 10.0%
* Willing to wear personal continuous glucose monitoring device (CGM)
* Willing to install and use CGM-linked app on personal smartphone with continuous access to WIFI or cellular data
* Able to read and write Korean as judged by investigator
* Willing to use medically acceptable contraception until end of study (sterile status, intrauterine device, or concurrent use of male/female barrier method with spermicide)
* Fully informed about the clinical trial and voluntarily consenting to participate

Exclusion Criteria:

* Type 1 diabetes mellitus
* Gestational diabetes mellitus
* History of pancreatectomy
* Continuous or intermittent insulin therapy for 7 days or more within 3 months
* Oral or IV steroid treatment within 1 month prior to informed consent
* Serious infection, surgery (scheduled or history), or severe trauma within 3 months prior to informed consent
* History of malignancy within 1 year prior to informed consent (except thyroid cancer)
* On hemodialysis or peritoneal dialysis or eGFR < 30 mL/min/1.73m2
* Unable to avoid the following concomitant medications, devices, or treatments during the study: CGM other than study device, X-ray/MRI/CT scans, radiofrequency thermal therapy, implantable devices such as pacemakers, immunosuppressants, steroids, IV vitamin preparations, cancer treatment, hemodialysis/peritoneal dialysis, insulin therapy
* Uncontrolled thyroid disease or clinically significant severe endocrine disorders (Cushing's syndrome, pheochromocytoma, etc.)
* Severe allergic reaction to skin adhesives (e.g., dyspnea, severe rash, edema)
* Whole blood donation within 60 days, apheresis within 30 days, or blood transfusion within 90 days prior to device application
* Judged by investigator as unable to handle continuous glucose monitoring device
* Pregnant or lactating women
* Planning pregnancy within 1 year
* Otherwise judged by investigator as inappropriate for participation in this clinical trial

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c from 3 to 6 months | At 6 months (V3)
  Non-inferiority comparison of the adjusted change in glycated hemoglobin A1c (HbA1c) from month 3 (V2, randomization visit) to month 6 (V3, end of study). The non-inferiority margin is set at 0.3%. The periodic use group will be considered non-inferior to the continuous use group if the lower bound of the 97.5% one-sided confidence interval for the difference in HbA1c change (periodic minus continuous) is greater than -0.3%.

SECONDARY OUTCOMES:
Change in HbA1c | At 6 months (V3)
  Adjusted change in glycated hemoglobin A1c (HbA1c) from month 3 to month 6, comparing periodic versus continuous CGM use groups.
Change in Blood Pressure | At 6 months (V3)
  Adjusted change in systolic and diastolic blood pressure from month 3 to month 6, comparing periodic versus continuous CGM use groups.
At 6 months (V3) | At 6 months (V3)
  Adjusted change in lipid parameters (LDL cholesterol, HDL cholesterol, total cholesterol, triglycerides) from month 3 to month 6, comparing periodic versus continuous CGM use groups.
Change in Body Weight | At 6 months (V3)
  Adjusted change in body weight (kg) from month 3 to month 6, comparing periodic versus continuous CGM use groups.
Change in HOMA-IR | At 6 months (V3)
  Adjusted change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) from month 3 to month 6, comparing periodic versus continuous CGM use groups.
Change in Diabetes Treatment Satisfaction (DTSQ) | At 6 months (V3)
  Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) score from month 3 to month 6, comparing periodic versus continuous CGM use groups. Higher scores indicate greater treatment satisfaction.
Change in Diabetes Self-Efficacy (K-DMSES) | At 6 months (V3)
  Change in Korean-Diabetes Management Self-Efficacy Scale (K-DMSES) score from month 3 to month 6, comparing periodic versus continuous CGM use groups. Higher scores indicate greater self-efficacy.
Change in Diabetes Self-Care Activities (SDSCA-K) | At 6 months (V3)
  Change in Summary of Diabetes Self-Care Activities Questionnaire-Korean (SDSCA-K) score from month 3 to month 6, comparing periodic versus continuous CGM use groups.
Time in Range 70-180 mg/dL (Non-inferiority) | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Non-inferiority comparison of percentage of time in glucose range 70-180 mg/dL between periodic and continuous CGM use groups. Non-inferiority margin is 6%.
Time in Range 70-180 mg/dL | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Percentage of time in glucose range 70-180 mg/dL, comparing periodic versus continuous CGM use groups.
Time in Tight Range 70-140 mg/dL | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Percentage of time in tight glucose range 70-140 mg/dL, comparing periodic versus continuous CGM use groups.
Time Above Range 180 mg/dL | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Percentage of time above glucose range (>180 mg/dL), comparing periodic versus continuous CGM use groups.
Time Above Range 250 mg/dL | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Percentage of time above glucose range (>250 mg/dL), comparing periodic versus continuous CGM use groups.
Time Below Range 70 mg/dL | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Percentage of time below glucose range (<70 mg/dL), comparing periodic versus continuous CGM use groups.
Time Below Range 54 mg/dL | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Percentage of time below glucose range (<54 mg/dL), comparing periodic versus continuous CGM use groups.
Glucose Standard Deviation (SD) | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Standard deviation of glucose levels, comparing periodic versus continuous CGM use groups.
Glucose Coefficient of Variation (CV) | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Coefficient of variation of glucose levels, comparing periodic versus continuous CGM use groups.
Mean Amplitude of Glycemic Excursions (MAGE) | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Mean amplitude of glycemic excursions, a measure of glucose variability, comparing periodic versus continuous CGM use groups.
Glucose Management Indicator (GMI) | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Glucose Management Indicator, an estimate of HbA1c derived from CGM data, comparing periodic versus continuous CGM use groups.
Mean Glucose | Combined period of 3.5-4 months, 4.5-5 months, and 5.5-6 months
  Mean glucose level (mg/dL), comparing periodic versus continuous CGM use groups

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in articles resulting from this study will be made available after deidentification. This includes data supporting primary and secondary outcomes, demographic information, and adverse event data. Data will be provided in a format suitable for secondary analysis while protecting participant privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data will be available beginning December 2028, approximately 24 months after the primary completion date. Data will be available for 5 years following initial availability. Supporting documents (protocol, SAP, CSR) will be made available at the same time.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for secondary analysis. Access will be granted at the discretion of the study investigators based on the scientific merit and feasibility of the proposed research.